CLINICAL TRIAL: NCT07118371
Title: Effects of Clamshell and Frog Pump Exercises on Pain, Range of Motion, and Functional Disability in Long-standing Sales Workers With Iliotibial Band Syndrome
Brief Title: Clamshell and Frog Pump Exercises on Pain, Range of Motion, and Functional Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/241/08/24
Record Dates: First submitted 2024-12-10; First posted 2025-08-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-10

CONDITIONS: Iliotibial Band Syndrome
Keywords: IT Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study will be single and assessor blinded. Participants will be masked about other groups but they will know what treatment they will be receiving or what exercises they will be doing. Principal investigator would also not be masked or blinded because investigator would be applying the techniques on participants of both group. So participant and and principal investigator cannot be blinded. Only assessor will be blinded and he will take outcome measures without knowing the problem and treatment techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamshell exercise (Experimental): The clamshell starts with lying on the side, with legs stacked and knees bent at a 45-degree angle. Rest the head on the lower arm and use the top arm to steady the frame. Hipbones are stacked on top of one another, as there is a tendency for the top hip to rock backward. Engage the abdominals by pulling your belly button in, as this will help to stabilize the spine and pelvis. Keeping the feet touching, raise the upper knee as high as they can without shifting the hips or pelvis. They don't move their lower leg off the floor. Pause, and then return the upper leg to the starting position on the ground. 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set.
  Interventions: Other: Clamshell exercise; Other: Frog pump exercises
- Frog pump exercises (Experimental): The Frog pump exercise will start with lying on your back, arms by sides, palms facing down. Alternatively, make fists with your hands, rest the elbows on the floor, and lift the fists so that your forearms are perpendicular to the floor. Then bend the knees and press the soles of the feet together so that the legs create a "frog legs" or "butterfly" shape. Pressing the outer edges of the feet against the floor, engage the core, and use the glutes to lift the hips. Make sure the shoulders and upper back remain anchored to the floor. Pause, then slowly lower the hips to the floor. . 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set.
  Interventions: Other: Clamshell exercise; Other: Frog pump exercises

INTERVENTIONS:
Other: Clamshell exercise — The clamshell starts with lying on the side, with legs stacked and knees bent at a 45-degree angle. Rest the head on the lower arm and use the top arm to steady the frame. Hipbones are stacked on top of one another, as there is a tendency for the top hip to rock backward. Engage the abdominals by pulling your belly button in, as this will help to stabilize the spine and pelvis. Keeping the feet touching, raise the upper knee as high as they can without shifting the hips or pelvis. They don't move their lower leg off the floor. Pause, and then return the upper leg to the starting position on the ground. 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set.
Other: Frog pump exercises — The Frog pump exercise will start with lying on your back, arms by sides, palms facing down. Alternatively, make fists with your hands, rest the elbows on the floor, and lift the fists so that your forearms are perpendicular to the floor. Then bend the knees and press the soles of the feet together so that the legs create a "frog legs" or "butterfly" shape. Pressing the outer edges of the feet against the floor, engage the core, and use the glutes to lift the hips. Make sure the shoulders and upper back remain anchored to the floor. Pause, then slowly lower the hips to the floor. . 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set.

SUMMARY:
The study will be randomized clinical trial. This study will be conducted at the University of Lahore Teaching Hospital, Lahore, Pakistan. A sample size of 92 will be randomly allocated into two experimental groups, (46 participants in each group), by the lottery method. All the screened and willing participants were randomly allocated into two groups (Group A: Experimental group / Clamshell exercise + Conservative management, Group B: Comparative Group / Frog pump exercises + Conservative management) by lottery method. The participants randomly allocated to Group A will receive conservative treatment along with clamshell exercise. The treatment will start with routine physiotherapy comprised of TENS (setting was in a conventional mode, with a frequency of 80 Hz and a pulse duration of 50-100 μs. The intensity of TENS current was set to produce a strong tingling sensation, but without pain.) A hot pack will be used for 10 minutes and stretching exercises for the whole body as a warm-up, before starting the main treatment regime for 15 minutes. The clamshell starts with lying on the side, with legs stacked and knees bent at a 45-degree angle. Group B will receive conservative treatment along with Frog pump exercise. The treatment will start with routine physiotherapy comprised of TENS (setting was in a conventional mode, with a frequency of 80 Hz and a pulse duration of 50-100 μs. The intensity of TENS current was set to produce a strong tingling sensation, but without pain.) A hot pack will be used for 10 minutes and stretching exercises for the whole body as a warm-up, before starting the main treatment regime for 15 minutes. The Frog pump exercise will start with lying on your back, arms by sides, palms facing down. Data will be assessed by the assessor at baseline, and at the end of the 12th week.

DETAILED DESCRIPTION:
Screening: All the participants will be assessed for the eligibility criteria. Patients fulfilling the eligibility criteria will be asked to sign the consent forms before entering them into the study.

Randomization and Allocation: All the screened and willing participants will be randomly allocated into two groups (Group A: Experimental group / Clamshell exercise + Conservative management, Group B: Comparative Group / Frog pump exercises + Conservative management) by lottery method.

Blinding: This study will be a single-blinded study in which the assessor will be blinded.

Intervention Group A: Experimental Group (Clamshell exercise + Conservative management) The participants randomly allocated to Group A will receive conservative treatment along with clamshell exercise. The treatment will start with routine physiotherapy comprised of TENS (setting was in a conventional mode, with a frequency of 80 Hz and a pulse duration of 50-100 μs. The intensity of TENS current was set to produce a strong tingling sensation, but without pain.) A hot pack will be used for 10 minutes and stretching exercises for the whole body as a warm-up, before starting the main treatment regime for 15 minutes. The clamshell starts with lying on the side, with legs stacked and knees bent at a 45-degree angle. Rest the head on the lower arm and use the top arm to steady the frame. Hipbones are stacked on top of one another, as there is a tendency for the top hip to rock backward. Engage the abdominals by pulling your belly button in, as this will help to stabilize the spine and pelvis. Keeping the feet touching, raise the upper knee as high as they can without shifting the hips or pelvis. They don't move their lower leg off the floor. Pause, and then return the upper leg to the starting position on the ground. 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set. The whole treatment session will start with 15 min warm-up and end with 5 min cool-down, delivered 3 times a week for 12 weeks yielding a total of 36 sessions within 3 months and the duration of each session will be of 35-45 minutes in Group A.

Group B: Comparative Group (Frog pump exercises + Conservative management) 19 Group B will receive conservative treatment along with Frog pump exercise. The treatment will start with routine physiotherapy comprised of TENS (setting was in a conventional mode, with a frequency of 80 Hz and a pulse duration of 50-100 μs. The intensity of TENS current was set to produce a strong tingling sensation, but without pain.) A hot pack will be used for 10 minutes and stretching exercises for the whole body as a warm-up, before starting the main treatment regime for 15 minutes. The Frog pump exercise will start with lying on your back, arms by sides, palms facing down. Alternatively, make fists with your hands, rest the elbows on the floor, and lift the fists so that your forearms are perpendicular to the floor. Then bend the knees and press the soles of the feet together so that the legs create a "frog legs" or "butterfly" shape. Pressing the outer edges of the feet against the floor, engage the core, and use the glutes to lift the hips. Make sure the shoulders and upper back remain anchored to the floor. Pause, then slowly lower the hips to the floor. . 20 reps will be done on each side. Each exercise will be performed in 3 sets of 10 repetitions with 1 minute of rest after every exercise set. The whole treatment session will start with 15 min warm-up and end with 5 min cool-down, delivered 3 times a week for 12 weeks yielding a total of 36 sessions within 3 months and the duration of each session will be of 35-45 minutes in Group B.

Outcome Variables:

1. Pain (Numeric Pain Rating Scale)
2. Range of Motion:(Goniometry)
3. Functional Disability (Lower Extremity Functional Scale (LEFS)) Data will be assessed by the assessor at baseline, and at the end of the 12th week.

ELIGIBILITY:
Inclusion Criteria:

* Both Males and Females
* Patients between the ages of 20 and 40
* Work shift (at least 4 hours a day) 5 times a week
* Positive Ober test
* Patients who have ITB band syndrome in one or both legs

Exclusion Criteria:

* Pregnant women
* Individuals have diseases or disorders that affect mobility.
* Recent Fractures of the lower limb
* Soft tissue injury of lower limb like ankle sprain etc.
* Severe systemic illnesses like COPD, Angina, or MI.
* Recent history of trauma
* Any psychiatric illness like panic disorders, obsessive-compulsive disorder, etc.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale) | 12 weeks
  Numeric rating scales consist of a series of numbers rating pain intensity, typically from 0 to 10 or 0 to 100, with 0 being "no pain" and 10 or 100 "the worst pain imaginable."
Goniometry) | 12 weeks
  A goniometer is an instrument that either measures an angle or allows an object to be rotated to a precise angular position.
Lower Extremity Functional Scale (LEFS) | 12 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ul Hassan, MS-MSK, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baik SM, Cynn HS, Shim JH, Lee JH, Shin AR, Lee KE. Effects of Log-Rolling Position on Hip-Abductor Muscle Activation During Side-Lying Hip-Abduction Exercise in Participants With Gluteus Medius Weakness. J Athl Train. 2021 Sep 1;56(9):945-951. doi: 10.4085/306-20. PMID 33150402
- [Background] Taddei UT, Matias AB, Duarte M, Sacco ICN. Foot Core Training to Prevent Running-Related Injuries: A Survival Analysis of a Single-Blind, Randomized Controlled Trial. Am J Sports Med. 2020 Dec;48(14):3610-3619. doi: 10.1177/0363546520969205. Epub 2020 Nov 6. PMID 33156692
- [Background] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Background] Bolia IK, Gammons P, Scholten DJ, Weber AE, Waterman BR. Operative Versus Nonoperative Management of Distal Iliotibial Band Syndrome-Where Do We Stand? A Systematic Review. Arthrosc Sports Med Rehabil. 2020 Jun 10;2(4):e399-e415. doi: 10.1016/j.asmr.2020.04.001. eCollection 2020 Aug. PMID 32875305
- [Background] Boonstra AM, Stewart RE, Koke AJ, Oosterwijk RF, Swaan JL, Schreurs KM, Schiphorst Preuper HR. Cut-Off Points for Mild, Moderate, and Severe Pain on the Numeric Rating Scale for Pain in Patients with Chronic Musculoskeletal Pain: Variability and Influence of Sex and Catastrophizing. Front Psychol. 2016 Sep 30;7:1466. doi: 10.3389/fpsyg.2016.01466. eCollection 2016. PMID 27746750
- [Background] Charles D, Rodgers C. A LITERATURE REVIEW AND CLINICAL COMMENTARY ON THE DEVELOPMENT OF ILIOTIBIAL BAND SYNDROME IN RUNNERS. Int J Sports Phys Ther. 2020 May;15(3):460-470. PMID 32566382
- [Background] Foch E, Aubol K, Milner CE. Relationship between iliotibial band syndrome and hip neuromechanics in women runners. Gait Posture. 2020 Mar;77:64-68. doi: 10.1016/j.gaitpost.2019.12.021. Epub 2020 Jan 20. PMID 31999979
- [Background] Geisler PR. Current Clinical Concepts: Synthesizing the Available Evidence for Improved Clinical Outcomes in Iliotibial Band Impingement Syndrome. J Athl Train. 2021 Aug 1;56(8):805-815. doi: 10.4085/1062-6050-548-19. Epub 2020 Dec 22. PMID 34375405
- [Background] Guerrero-Tapia H, Martin-Baeza R, Cuesta-Barriuso R. Effectiveness of Abdominal and Gluteus Medius Training in Lumbo-Pelvic Stability and Adductor Strength in Female Soccer Players. A Randomized Controlled Study. Int J Environ Res Public Health. 2021 Feb 5;18(4):1528. doi: 10.3390/ijerph18041528. PMID 33562743
- [Background] Hong JH, Kim JS. Diagnosis of iliotibial band friction syndrome and ultrasound guided steroid injection. Korean J Pain. 2013 Oct;26(4):387-91. doi: 10.3344/kjp.2013.26.4.387. Epub 2013 Oct 2. PMID 24156006